CLINICAL TRIAL: NCT03241953
Title: COMPARISION OF DIFFERENT TREATMENT METHODS OF PERI-IMPLANTITIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, ELİF ONCU, Asist.Prof.Dr., Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014-08
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Peri-Implantitis; Periodontal Diseases
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- debridement made by ultrasonic tips (Experimental): mechanical debridement made by ultrasonic polyetheretherketone coated tips developed for implant surface and combined air-flow debridement
  Interventions: Procedure: Periodontal surgery
- implants were debrided with standard plastic curettes (Active Comparator): dental implants were debrided with standard plastic curettes, debridement made by combined klorhegsidin rinse
  Interventions: Procedure: Periodontal surgery

INTERVENTIONS:
Procedure: Periodontal surgery — A total of forty dental implants were debrided with either ultrasonic instruments (test, n=20) or plastic scaler (control, n=20). Gingival recession depth (RD), keratinized tissue width (KTW), probing depth (PD), Gingival Index (GI) were evaluated at baseline and after 6 months. CBCT radiographs were used to evaluate peri-implant bone loss. Supportive and nonsurgical periodontal therapies were firstly consulted to reduce the inflammation, occurring due to the surgical treatments of the defects. The formation of bacterial biofilm on implant surfaces was removed by ultrasonic scaler and air polishing

SUMMARY:
In this randomized, controlled study, 18 patients with peri-implantitis were included. A total of forty dental implants were debrided with either ultrasonic instruments (test, n=20) or plastic scaler (control, n=20). Gingival recession depth (RD), keratinized tissue width (KTW), probing depth (PD), Gingival Index (GI) were evaluated at baseline and after 6 months. CBCT radiographs were used to evaluate peri-implant bone loss. Supportive and nonsurgical periodontal therapies were firstly consulted to reduce the inflammation, occurring due to the surgical treatments of the defects. The formation of bacterial biofilm on implant surfaces was removed by ultrasonic scaler and air polishing using abrasive powders or conventional plastic scaler with klorhegsidin combination.

DETAILED DESCRIPTION:
Subject selection 18 systemically healthy patients, who applied to the Department of Periodontology, Necmettin Erbakan University and whose at least 1 dental implant was diagnosed by peri-implantitis and who has never taken peri-implantitis therapy, were included in the study. All patients were informed about the study and given informed consent form, and only volunteers were included. The research was conducted in accordance with the principles outlined in the Declaration of Helsinki. This prospective clinical study was approved by the Research Ethics Committee of Necmettin Erbakan University.

The patients, who were systemically and periodontally healthy and free of parafunctional habits like bruxism, and didn't have any kind of periodontal therapy within the previous year and had implants for at least 5 years, were included in the study. In addition, the inclusion criteria were as follows: having pocket depth over 5mm in implants diagnosed by peri-implantitis (Figure 1), having no mobility, having bone loss in implant site that is needed for augmentation(Figure 2). The patients with chronic bronchitis or asthma and major systemic illnesses (i.e. diabetes mellitus, cancer, HIV, bone metabolic diseases or disorders that compromise wound healing, radiation or immunosuppressive therapy) and those who had taken antibiotics, anti-inflammatory drugs or other medication within the previous 28 days were excluded in the study.

18 patients (mean age 52 years) diagnosed by peri- implantitis were included in this randomized and controlled study. A total of forty dental implants were debrided with either standard plastic curettes, debridement made by combined klorhegsidin rinse(control, n=20) or mechanical debridement made by ultrasonic polyetheretherketone coated tips developed for implant surface and combined air-flow debridement (test, n=20).

Clinical Measurements The clinical parameters given below were observed on six sites of all implants: Plaque Index (PlI; Silness & Lo€e 1964), PD, Bleeding upon Probing (BOP) and Gingival Recession (RD; gingival margin location measuremant cemento- enamel junction to Gingival marjin).

On six sites of all implants, the following clinical parameters were recorded: Plaque Index (PlI; Silness & Lo€e 1964), PD, Bleeding on Probing (BOP) and Gingival Recession (RD; gingival margin location measuremant cemento- enamel junction to Gingival marjin).

Keratinized tissue width (KTW) was measured at buccal midpoint of implants. Bone loss volume was recorded on con-beam computed tomographs (CBCT) by measuring the distance from bone implant abutment placement to alveolar bone level. All measurements were taken at the beginning. As we didn't perform any regenerative operations and didn't want the patients to be subjected to X-rays again, no more tomographs were taken.

Phase I Periodontal Therapy Upon the recordings, all patients were given Phase 1 periodontal therapy and informed about hygiene control. Prior to surgical operation, professional supragingival and subgingival debridement was performed during 2 or 4 appointments. The patients with a good level of oral hygiene were included in the study. Oral hygiene controls were performed in the first, third and sixth months prior to and after operations. Occlusion controls of all implant supported dental prosthesis were performed, and if present, extreme contacts were removed.

Phase II Periodontal Therapy 4 weeks after the initial periodontal treatments, for the treatment of the sites with pocket depth deeper than 5mm, flap operation was performed to achieve a direct reach to implant surfaces. Around affected implants, intrasulcular incisions were performed and mucoperiostal flaps with full thickness were raised both buccally and palatally. Implant surface decontamination is performed using with either plastic curettes or ultrasonic scaler (Figure 3); In control group, plastic curettes (Hue-Friedy Co., Chicago, IL, USA) were used for debridement and implant surfaces were decontaminated by klorhegsidin solution. In test group, sub-gingival operations with ultrasonic scaler was for nearly 20s per site (EMS Master Piezon LED, implant care system, Nyon, Switzerland). A special design disposable thermoplastic elastomer nozzle (Perio-flow Nozzle EMS Electro Medical Systems, Nyon, Sweden.), which horizontally gives out the glycine powder, was utilized.

The hand-device (Air-Flows EL-308/A; EMS Electro Medical Systems, Nyon, Sweden) was used in a circular motion, from coronal to apical, parallel to the implant surface in a noncontact mode. The operation period time at each aspect (i.e. mesial, distal, vestibular and oral) was limited to 5 s, as suggested by the manufacturer 35. The nozzle was moved with a circumferential movement around the implant to cover the entire exposed implant surface (36).

After the debriding of implant surfaces the flap was sutured by 4-0 vicryl. After the operation, for antimicrobial treatment chlorhexidine was used for 10 days. The sutures were removed 10 days after the operation and post-operative controls were performed. The patients were invited to the followups in the first, third and sixth month after the operation. Clinical and radiographic measurements were repeated every six months

ELIGIBILITY:
Inclusion Criteria:

- The patients, who were systemically and periodontally healthy and free of parafunctional habits like bruxism, and didn't have any kind of periodontal therapy within the previous year and had implants for at least 5 years, were included in the study.

Exclusion Criteria:

* The patients with chronic bronchitis or asthma and major systemic illnesses (i.e. diabetes mellitus, cancer, HIV, bone metabolic diseases or disorders that compromise wound healing, radiation or immunosuppressive therapy) and those who had taken antibiotics, anti-inflammatory drugs or other medication within the previous 28 days were excluded in the study.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2014-04-23 (Actual); Primary Completion 2016-11-20 (Actual); Study Completion 2016-12-22 (Actual)

PRIMARY OUTCOMES:
Treatment results | one year
  It was found in the study that the combined air-flow debridement and the mechanical debridement performed by using ultrasonic polyetheretherketone-coated tips developed for implant surface debridement in peri-implantitis therapy were better at decreasing the level of periodontal pocket depth than plastic curettes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/21770995
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/21251076